CLINICAL TRIAL: NCT03475329
Title: Adenoidectomy With Bilateral Partial Tonsillectomy Versus Adenoidectomy With Unilateral Complete Tonsillectomy in Treatment of Children With Obstructive Sleep-Disordered Breathing :Acomparative Study
Brief Title: Adeno-tonsillectomy in Treatment of Obstructive Sleep Apnea
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Christina Farag Zaki, the principal investigator, Assiut University
Other Study IDs: AITOOSA
Record Dates: First submitted 2018-03-12; First posted 2018-03-23 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Obstructive Sleep Disordered Breathing
Keywords: pediatric obstructive sleep disordered breathing-partial tonsillectomy -unilateral complete tonsillectomy -adenoidectomy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- adenoidectomy with bilateral partial tonsillectomy
  Interventions: Other: adenotonsillectomy
- adenoidectomy with complete unilateral tonsillectomy
  Interventions: Other: adenotonsillectomy

INTERVENTIONS:
Other: adenotonsillectomy — adenoidectomy with bilateral tonsillectomy versus adenoidectomy with unilateral complete tonsillectomy

SUMMARY:
The aim of the study is to evaluate adenoidectomy with bilateral partial tonsillectomy compared with adenoidectomy with classical unilateral complete tonsillectomy for management of pediatric Obstructive Sleep-Disordered Breathing (OSDB) in terms of efficacy of the technique and reducing postoperative complications.

DETAILED DESCRIPTION:
Tonsillectomy is one of commonly performed pediatric otorhinolaryngology surgeries.

The two main indications of tonsillectomy in children include recurrent tonsillitis and Obstructive Sleep-Disordered Breathing (OSDB); including obstructive sleep apnea and upper airway resistance syndrome.

Total tonsillectomy means total removal of the tonsillar tissue with the tonsillar capsule. The main drawbacks of tonsillectomy are the potential for serious postoperative bleeding, postoperative pain, eating and drinking difficulties, and reduced immune function in the early stages after the operation. Partial tonsillectomy (intracapsular tonsillectomy, subtotal tonsillectomy) means subtotal removal of tonsillar tissue, leaving a margin of tissue on the tonsillar capsule . In contrast to complete tonsil removal, Partial tonsillectomy does not violate the capsule, and leaves lymphoid tissue as a protective tissue on the pharyngeal muscle layer thus preserving of the connective tissue capsule and pharyngeal muscles. This diminishes the direct and indirect trauma during an intraoperative procedure and the inflammation due to secondary infection during the postoperative period. Recently, children with OSDB have benefited from the less invasive partial tonsillectomy with less pain, equivalent or easier recovery, better food intake, and maintain the immunological function of the tonsils, while being as effective as tonsillectomy for resolving upper-airway obstructive symptoms.

Many studies have evaluated the outcomes of the two techniques, but uncertainty remains with regard to the efficacy, complications and long term outcomes. Some studies have reported the recurrence of obstructive symptoms due to regrowth of the remaining tonsillar tissue. Thus, it is important to evaluate Partial tonsillectomy comprehensively, especially paying attention to short-term and long-term results.

Over the last years, unilateral complete tonsillectomy (usually combined with adenoidectomy) was the most commonly utilized procedure for treatment of pediatric obstructive sleep-disordered breathing below the age of four years old in Otorhinolaryngology Department, Assiut University

ELIGIBILITY:
Inclusion Criteria:

* • Age: 1-3 yeas.

  * Diagnosed to have Obstructive Sleep-Disordered Breathing (OSDB) due to adenotonsillar enlargement confirmed by flexible nasoendoscopic assessment.

Exclusion Criteria:

* • Any associated medical comorbidity that contraindicates general anesthesia.

  * Children having other causes for OSDB (e.g. obesity, Down syndrome, craniofacial abnormalities, neuromuscular disorders, sickle cell disease, or mucopolysaccharidoses).
  * Refusal of enrollment in the research by care givers.

Ages: 1 Year to 3 Years | Sex: All
Age Groups: Child
Study Population: The study will be conducted on Otorhinolaryngology Department, Assiut University Hospital.The study will be carried on 60 consecutive cases.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-01-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain assessed by cries scale | two weeks
  The CRIES scale is used for infants > than or = 38 weeks of gestation. Characteristics of crying, oxygen requirement, changes in vital signs, facial expression, and sleep state are scored. A maximal score of 10 is possible. If the CRIES score is > 4, further pain assessment should be undertaken, and analgesic administration is indicated for a score of 6 or higher.

CONTACTS AND LOCATIONS:
Locations (1):
- Assuit, Asyut, Egypt